CLINICAL TRIAL: NCT05828667
Title: The STandard Versus ImAging SuBstrate Aided Ablation in Severe Left VEntricular
Brief Title: The STandard Versus ImAging SuBstrate Aided Ablation in Severe Left VEntricular Dysfunction VT.
Acronym: STABLE-VT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Potential protocol modifications are pending, and enrollment has been challenging.
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 851281
Record Dates: First submitted 2023-03-06; First posted 2023-04-25 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: A randomized controlled non-blinded prospective single-center study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care Arm (No Intervention): Standard of care procedural steps per respective institution and attending physician's clinical practice.
- Imaging-aided VT ablation (Experimental): For subjects assigned to the imaging-aided VT ablation arm, CT and/or c-MRI derived myocardial scar will be merged with 3D electroanatomical mapping (EAM) prior to the ablation to allow for readily localization and characterization of VT substrates and potential re-entry circuits to be ablated. This integrated mapping of VT substrates sites to be ablated will be given to the electrophysiologist prior to the ablation.
  Interventions: Other: Incorporation of CT and/or c-MRI derived myocardial scar with 3D electroanatomical mapping (EAM).

INTERVENTIONS:
Other: Incorporation of CT and/or c-MRI derived myocardial scar with 3D electroanatomical mapping (EAM). — CT and/or c-MRI derived myocardial scar will be merged with 3D electroanatomical mapping (EAM) prior to the ablation to allow for readily localization and characterization of VT substrates and potential re-entry circuits to be ablated. This is done with the intent to limit the repeated number of inductions and prolonged point-by-point voltage mapping that often result in hemodynamic instability.
  Arms: Imaging-aided VT ablation

SUMMARY:
The STABLE-VT trial aims to determine the safety profile and clinical efficacy of a modified approach to ventricular tachycardia (VT) ablation that integrates myocardial scar as visualized on cardiac magnetic resonance (c-MRI) or CT into electroanatomical mapping (EAM) for VT ablation.

DETAILED DESCRIPTION:
The STABLE-VT trial aims to integrate myocardial scar as visualized on cardiac magnetic resonance (c-MRI) or CT into electroanatomical mapping (EAM) for VT ablation. Particularly, we will compare the procedural safety, and acute and long-term clinical efficacy of this imaging-aided VT ablation protocol to standard of care.

Our hypothesis is that patients with ventricular tachycardia (VT) and severe LV dysfunction randomized to this imaging-aided protocol will have shorter procedure duration, improved procedural hemodynamic stability, fewer acute major adverse cardiovascular events (MACE), less need for mechanical support, comparable freedom from VT at noninvasive programmed stimulation (NIPS) sub-acutely after the procedure, and at two-year follow-up compared to standard ablation approach. Herein, our outcomes of interest will be captured during the two years following as part of regular standard of care follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* Patients (>18 years old) diagnosed with severely reduced ejection fraction defined as EF≤25% or EF≤ 35% with concurrent NYHA class III/IV heart failure symptoms and/or at least one previous heart failure hospitalization in the previous 6 months) who are referred for VT ablation.
* Patients with moderate to severe RV dysfunction diagnosed on most recent imaging (echo/c-MRI).
* Patients with must have undergone the imaging (c-MRI and/or CT) required for the investigational VT approach to qualify for participation.

Exclusion Criteria:

* Patients in whom Impella/ECMO or anesthesia is indicated prior to or at presentation to the EP lab.
* Patients for whom an informed consent cannot be obtained.
* Patients who are found to be pregnant using detection of human chorionic gonadotropin (hcg) as done as part of standard of care, will be excluded.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiovascular events (MACE) | during hospital stay following ablation procedure, up to 1 week
  Incidence of major adverse cardiac events, which are cardiovascular death, myocardial infarction, stroke/TIA
Number of Participants Requiring Mechanical circulatory support use | During the procedure, 24-48 hours after the ablation procedure
  Incidence of mechanical circulatory support (e.g., extra corporeal membrane oxygenation, Impella, LVAD or transplant) use
Number of Participants Requiring Inotropic support use | During the procedure, 24-48 hours after the ablation procedure
  Incidence of inotropic and vasoactive agents use
Number of Participants With Clinically Significant Pericardial Effusion | During the procedure, up to 24 hours after the ablation procedure
  Assessing clinically significant pericardial effusion causing hemodynamic instability
Number of Participants With Acute kidney injury | During procedure, up to 24-48 hours after the ablation procedure
  Acute kidney injury (≥50% within 48 hours of the start of the procedure)
Number of Participants Requiring intubation | During procedure, 24 hours after the ablation procedure
  Need for intubation

SECONDARY OUTCOMES:
Experimental procedural duration | During procedure
  Experimental procedural duration
noninvasive programmed stimulation (NIPS) sub-acutely after the procedure | 24-48 hours after the procedure.
  comparable freedom from VT at noninvasive programmed stimulation (NIPS) sub-acutely after the procedure and at two-year follow-up.
Mean and peak procedural lactate level | During procedure
  Mean and peak procedural lactate level
Cumulative procedural inotropic support use | During procedure, 24-48 hours after the ablation procedure
  Cumulative procedural inotropic support use
Hospital stay length following the procedure | Periprocedural hospital stay length, up to 2 weeks
  Hospital stay length following the procedure
Time to ventricular tachycardia (VT) | 1 year
  Time to recurrent VT or censoring at 1 year (detection 10 bpm < rate of slowest VT)
Antiarrhythmic Drugs requirement | Through study completion, an average of 1 year
  Antiarrhythmic Drugs requirement following the procedure
Left ventricular ejection fraction (LVEF) | 6 months after the study
  Change in LVEF at 6 months at regular clinic follow-ups following the procedure
Left ventricular end-diastolic volume (EDV) | 6 months after the study
  Change in EDV at 6 months at regular clinic follow-ups following the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of The University Of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bogun FM, Desjardins B, Good E, Gupta S, Crawford T, Oral H, Ebinger M, Pelosi F, Chugh A, Jongnarangsin K, Morady F. Delayed-enhanced magnetic resonance imaging in nonischemic cardiomyopathy: utility for identifying the ventricular arrhythmia substrate. J Am Coll Cardiol. 2009 Mar 31;53(13):1138-45. doi: 10.1016/j.jacc.2008.11.052. PMID 19324259
- [Background] Wijnmaalen AP, van der Geest RJ, van Huls van Taxis CF, Siebelink HM, Kroft LJ, Bax JJ, Reiber JH, Schalij MJ, Zeppenfeld K. Head-to-head comparison of contrast-enhanced magnetic resonance imaging and electroanatomical voltage mapping to assess post-infarct scar characteristics in patients with ventricular tachycardias: real-time image integration and reversed registration. Eur Heart J. 2011 Jan;32(1):104-14. doi: 10.1093/eurheartj/ehq345. Epub 2010 Sep 23. PMID 20864488
- [Background] Andreu D, Berruezo A, Ortiz-Perez JT, Silva E, Mont L, Borras R, de Caralt TM, Perea RJ, Fernandez-Armenta J, Zeljko H, Brugada J. Integration of 3D electroanatomic maps and magnetic resonance scar characterization into the navigation system to guide ventricular tachycardia ablation. Circ Arrhythm Electrophysiol. 2011 Oct;4(5):674-83. doi: 10.1161/CIRCEP.111.961946. Epub 2011 Aug 31. PMID 21880674
- [Background] Komatsu Y, Cochet H, Jadidi A, Sacher F, Shah A, Derval N, Scherr D, Pascale P, Roten L, Denis A, Ramoul K, Miyazaki S, Daly M, Riffaud M, Sermesant M, Relan J, Ayache N, Kim S, Montaudon M, Laurent F, Hocini M, Haissaguerre M, Jais P. Regional myocardial wall thinning at multidetector computed tomography correlates to arrhythmogenic substrate in postinfarction ventricular tachycardia: assessment of structural and electrical substrate. Circ Arrhythm Electrophysiol. 2013 Apr;6(2):342-50. doi: 10.1161/CIRCEP.112.000191. Epub 2013 Mar 10. PMID 23476043
- [Background] Liang JJ, Muser D, Santangeli P. Ventricular Tachycardia Ablation Clinical Trials. Card Electrophysiol Clin. 2017 Mar;9(1):153-165. doi: 10.1016/j.ccep.2016.10.012. Epub 2016 Dec 24. PMID 28167083
- [Background] Santangeli P, Muser D, Maeda S, Filtz A, Zado ES, Frankel DS, Dixit S, Epstein AE, Callans DJ, Marchlinski FE. Comparative effectiveness of antiarrhythmic drugs and catheter ablation for the prevention of recurrent ventricular tachycardia in patients with implantable cardioverter-defibrillators: A systematic review and meta-analysis of randomized controlled trials. Heart Rhythm. 2016 Jul;13(7):1552-9. doi: 10.1016/j.hrthm.2016.03.004. Epub 2016 Mar 4. PMID 26961297
- [Background] Liang JJ, Santangeli P, Callans DJ. Long-term Outcomes of Ventricular Tachycardia Ablation in Different Types of Structural Heart Disease. Arrhythm Electrophysiol Rev. 2015 Dec;4(3):177-83. doi: 10.15420/aer.2015.4.3.177. Epub 2015 Dec 1. PMID 26835122
- [Background] Santangeli P, Muser D, Zado ES, Magnani S, Khetpal S, Hutchinson MD, Supple G, Frankel DS, Garcia FC, Bala R, Riley MP, Lin D, Rame JE, Schaller R, Dixit S, Marchlinski FE, Callans DJ. Acute hemodynamic decompensation during catheter ablation of scar-related ventricular tachycardia: incidence, predictors, and impact on mortality. Circ Arrhythm Electrophysiol. 2015 Feb;8(1):68-75. doi: 10.1161/CIRCEP.114.002155. Epub 2014 Dec 9. PMID 25491601
- [Background] Santangeli P, Frankel DS, Tung R, Vaseghi M, Sauer WH, Tzou WS, Mathuria N, Nakahara S, Dickfeldt TM, Lakkireddy D, Bunch TJ, Di Biase L, Natale A, Tholakanahalli V, Tedrow UB, Kumar S, Stevenson WG, Della Bella P, Shivkumar K, Marchlinski FE, Callans DJ; International VT Ablation Center Collaborative Group. Early Mortality After Catheter Ablation of Ventricular Tachycardia in Patients With Structural Heart Disease. J Am Coll Cardiol. 2017 May 2;69(17):2105-2115. doi: 10.1016/j.jacc.2017.02.044. PMID 28449770
- [Background] Tzou WS, Tung R, Frankel DS, Vaseghi M, Bunch TJ, Di Biase L, Tholakanahalli VN, Lakkireddy D, Dickfeld T, Saliaris A, Weiss JP, Mathuria N, Tedrow U, Afzal MR, Vergara P, Nagashima K, Patel M, Nakahara S, Vakil K, Burkhardt JD, Tseng CH, Natale A, Shivkumar K, Callans DJ, Stevenson WG, Della Bella P, Marchlinski FE, Sauer WH. Ventricular Tachycardia Ablation in Severe Heart Failure: An International Ventricular Tachycardia Ablation Center Collaboration Analysis. Circ Arrhythm Electrophysiol. 2017 Jan;10(1):e004494. doi: 10.1161/CIRCEP.116.004494. PMID 28082527
- [Background] Zghaib T, Ipek EG, Hansford R, Ashikaga H, Berger RD, Marine JE, Spragg DD, Tandri H, Zimmerman SL, Halperin H, Brancato S, Calkins H, Henrikson C, Nazarian S. Standard Ablation Versus Magnetic Resonance Imaging-Guided Ablation in the Treatment of Ventricular Tachycardia. Circ Arrhythm Electrophysiol. 2018 Jan;11(1):e005973. doi: 10.1161/CIRCEP.117.005973. No abstract available. PMID 29330333